CLINICAL TRIAL: NCT03780777
Title: Removing Home Hazards for Older Adults in Affordable Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: US Department of Housing and Urban Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201811108; MOHHU0040-17 (Other Grant/Funding Number: U.S. Department of Housing and Urban Development)
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Accidental Fall
Keywords: older adult falls; home hazards; home barriers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home Hazard Removal Group (Experimental): A tailored home-modification (home-hazard removal) intervention for residents with a high fall risk, delivered in the home by occupational therapists over one to two visits and with a booster session at three months.
  Interventions: Behavioral: Home Hazard Removal

INTERVENTIONS:
Behavioral: Home Hazard Removal — Removal of home barriers or hazards

SUMMARY:
The investigators will conduct a hybrid effectiveness/implementation trial to simultaneously establish the effectiveness of home hazard removal in affordable housing in order to reduce falls, and conduct a process evaluation of how the intervention works in the context of low-income senior apartments.

DETAILED DESCRIPTION:
The investigators, in collaboration with the community partner, will offer the program to all building residents in select low-income senior apartments. The eligibility criteria include a self-report of one or more falls in the preceding 12 months, a fear of falling, or unsteadiness while standing or walking. The investigators will screen residents and determine their risk for falling. Residents who are high risk will be referred to licensed occupational therapy practitioners for baseline assessments and home hazard removal. Residents will be re-assessed at 3 months. All assessments will be conducted in the residents' apartment buildings. Outcomes (falls, program evaluation) will be collected by our community partner.

ELIGIBILITY:
Inclusion Criteria:

* Residents who live in any of the eligible section 202 low-income senior apartment units managed by our community partner

Exclusion Criteria:

* Individuals who do not reside in any of the eligible units

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Resident enrollment in home hazard removal intervention | 609 days
  Participation measured by percentage of eligible building residents enrolled
Program fidelity | 609 days
  Visit-by-visit checklist and calculation of the dose of the intervention received (number of minutes delivered)

SECONDARY OUTCOMES:
Number of falls | 609 days
  Prospective monthly reporting of falls using an automated phone system
Cost per fall prevented | 609 days
  Final prescription and invoice (materials)
Adherence to home hazard removal intervention recommendations | 609 days
  Recommendations used/total at 3 months or cause of abandonment

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No